CLINICAL TRIAL: NCT02016794
Title: A Focused Registry on Anterior Cervical Interbody Spacer Procedures in Patients With Cervical Spine Degeneration
Brief Title: A Focused Registry on Anterior Cervical Interbody Spacer ACIS
Acronym: ACIS
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FR_ACIS
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Degenerative Cervical Spine
Keywords: cervical; interbody; spacer; degenerative; pain; neck; decompression; fusion; implant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients suffering from degenerative cervical condition that requires anterior decompression and fusion in a single or multiple levels

SUMMARY:
Degenerative cervical spine conditions lead to chronic neck and arm pain. Surgical treatment may require anterior decompression and fusion, which usually is established with a cage implant. The Anterior Cervical Interbody Spacer (ACIS) is such a cage.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Degenerative cervical condition that requires anterior decompression and fusion in a single or multiple levels
* Degenerative cervical disc disease C3 through Th1 or
* Ruptured and herniated discs C3 through Th1
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the registry according to the registry plan (RP)
* Signed and dated IRB / EC-approved written informed consent

Exclusion Criteria:

* Spinal tumor
* Osteoporosis
* Cervical trauma and instability
* Any not medically managed severe systemic disease (ie. infection)
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the registry period
* Prisoner
* Participation in any other medical device or medicinal product clinical investigation or registry within the previous month that could influence the results of the present registry

Intraoperative exclusion criteria:

* Intraoperative decision to use implants other than the device under investigation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for degenerative cervical condition that requires anterior decompression and fusion in a single or multiple levels
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Effect of neck pain on everyday life measured by the Neck Disability Index (NDI). | 6 months

SECONDARY OUTCOMES:
Pain | Baseline; 1-2days; 6 weeks; 6 months
  Numeric Rating Scale
Handling details | Intraoperative
  easiness of using ACIS, overall satisfaction with ACIS, time of surgery
Length of Hospital Stay | Expected average of 5 days
  From the day of the surgery until the day of discharge
Adverse Events | Intra and post operative

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Klina, Brasschaat
  - AZ Sint Maarten, Duffel